CLINICAL TRIAL: NCT03083808
Title: A Phase II Trial of Chemotherapy Plus Pembrolizumab in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Previously Treated With PD-1 or PD-L1 Inhibitor: Big Ten Cancer Research Consortium BTCRC-LUN15-029
Brief Title: Phase II Trial of Continuation Therapy in Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Greg Durm, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Greg Durm, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-LUN15-029
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: PD-1; PD-L1 Inhibitor; Pembrolizumab; Docetaxel; Pemetrexed; Gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab 200mg IV every 21 days (Experimental): Patients who have been treated with a PD-1 or PD-L1 inhibitor and experienced a PFS of ≥3 months will be enrolled within 6 weeks of last dose of PD-1 or PD-L1 inhibitor. On Day 1 of each 3-week cycle, subjects will first receive pembrolizumab at a dose of 200mg IV every three weeks in combination with chemotherapy. Partner chemotherapy will be either gemcitabine 1000mg/m^2 IV D1 and D8 every three weeks, docetaxel 75mg/m^2 IV D1 every three weeks, or pemetrexed 500mg/m^2 IV D1 every 3 weeks (pemetrexed for non-squamous histologies only). Subjects will continue to receive this combination until progression or intolerable toxicity.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg IV every 21 days
  +
  Physician's choice chemotherapy with one of the following every 21 days:
  * Docetaxel 75mg/m2 IV
  * Pemetrexed 500mg/m2 IV (non-squamous only)
  * Gemcitabine 1000mg/m2 IV on days 1 and 8
  Other Names: Keytruda®; MK-3475

SUMMARY:
This is a single-arm phase II study of continuation immunotherapy with pembrolizumab following initial benefit (CR, PR, or SD ≥ 3 months) with a PD-1 or PD-L1 inhibitor.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Patients who have been treated with a PD-1 or PD-L1 inhibitor and experienced a PFS of ≥3 months will be enrolled within 6 weeks of last dose of PD-1 or PD-L1 inhibitor. On Day 1 of each 3-week cycle, subjects will first receive pembrolizumab at a dose of 200mg IV every three weeks in combination with chemotherapy. Partner chemotherapy will be either gemcitabine 1000mg/m2 IV D1 and D8 every three weeks, docetaxel 75mg/m2 IV D1 every three weeks, or pemetrexed 500mg/m2 IV D1 every 3 weeks (pemetrexed for non-squamous histologies only). Subjects will continue to receive this combination until progression or intolerable toxicity.

Administration Sequence: First Sequence

- Pembrolizumab 200mg IV on Day 1 (cycle = 21 days)

Administration Sequence: Second Sequence

* Gemcitabine 1000mg/m^2 IV on Days 1,8 (cycle = 21 days)
* Docetaxel 75mg/^2 IV on Days 1,8 (cycle = 21 days)
* Pemetrexed 500mg/m^2 IV on Day 1 (cycle -= 21 days)

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of protected health information.
* Age ≥ 18 years at the time of consent.
* Histological or cytological evidence of stage IV NSCLC (any histology)
* Subjects must have progressed on or after previous platinum-based chemotherapy. Chemotherapy may have previously been given with a PD-1 or PD-L1 inhibitor. Subjects must have also progressed on or after receiving any PD-1 or PD-L1 inhibitor (including pembrolizumab) as their most recent therapy and must have had at least a 3-month PFS on this therapy.
* Subjects must be enrolled on the trial within 6 weeks of their last infusion of PD-1 or PD-L1 inhibitor therapy.
* Subjects whose tumors harbor a mutation in EGFR exon 19 or 21 or have gene rearrangements in ALK or ROS1 must have already been treated with standard targeted therapies. NOTE: Subjects must also have progressed on or after platinum-containing combination chemotherapy.
* ECOG Performance Status of 0 or 1 within 28 days prior to registration for protocol therapy.
* Must be fit enough to receive next-line chemotherapy (either gemcitabine, docetaxel, or pemetrexed [non-squamous only]) according to the discretion of the treating physician.
* Adequate laboratory values obtained within 28 days prior to registration for protocol therapy.
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test within 7 days prior to study registration and/or within 72 hours of first dose of study drugs. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Women of childbearing potential must be willing to use two methods of contraception or abstain from heterosexual activity from the point of registration through 120 days after the last dose of study drug.
* Male subjects capable of fathering a child must agree to use an adequate method of contraception starting with the first dose of the study drug through 120 days after the last dose of the study drug.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Active central nervous system (CNS) metastases. NOTE: Subjects who are symptomatic or have not undergone prior brain imaging must undergo a head computed tomography (CT) scan or brain MRI within 28 days prior to registration to exclude brain metastases.
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy with the exception of PD-1 or PD-L1 inhibitors.
* No active second cancers with the exception of localized non-melanoma skin cancer, in-situ cervical or in-situ bladder cancer.
* Evidence of active autoimmune disease requiring systemic treatment within the past 90 days or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* History of (non-infectious) pneumonitis requiring treatment with corticosteroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* History of an immune-related toxicity requiring treatment with corticosteroids during prior PD-1/ PD-L1 inhibitor treatment.
* Diagnosis of immunodeficiency or is receiving chronic systemic corticosteroid therapy or other immunosuppressive therapy (excludes inhaled corticosteroids) within 7 days of study registration.
* History of psychiatric illness or social situations that would limit compliance with study requirements.
* Clinically active infection (≥ Grade 2) as judged by the site investigator.
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C. NOTE: HIV, HBV or HCV testing is not required.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
* Known history of active TB (Bacillus Tuberculosis).
* History of hypersensitivity to pembrolizumab, docetaxel, gemcitabine, pemetrexed or any of their excipients.
* Has received a live vaccine within 30 days prior to planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Durm, M.D., Study Chair — Big Ten Cancer Research Consortium
Locations (5):
- United States (5):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospital Clinics, Iowa City, Iowa
  - University of Minnesota Medcical Center, Minneapolis, Minnesota
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab 200mg IV Every 21 Days: Patients who have been treated with a PD-1 or PD-L1 inhibitor and experienced a PFS of ≥3 months will be enrolled within 6 weeks of last dose of PD-1 or PD-L1 inhibitor. On Day 1 of each 3-week cycle, subjects will first receive pembrolizumab at a dose of 200mg IV every three weeks in combination with chemotherapy. Partner chemotherapy will be either gemcitabine 1000mg/m^2 IV D1 and D8 every three weeks, docetaxel 75mg/m^2 IV D1 every three weeks, or pemetrexed 500mg/m^2 IV D1 every 3 weeks (pemetrexed for non-squamous histologies only). Subjects will continue to receive this combination until progression or intolerable toxicity.
  Pembrolizumab: Pembrolizumab 200mg IV every 21 days
  +
  Physician's choice chemotherapy with one of the following every 21 days:
  * Docetaxel 75mg/m2 IV
  * Pemetrexed 500mg/m2 IV (non-squamous only)
  * Gemcitabine 1000mg/m2 IV on days 1 and 8
Period: Overall Study
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 63 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 35
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 26
  Squamous cell carcinoma | 7
  Non-small cell, not otherwise specified | 2
Smoking Status [Count of Participants; unit: Participants]
  Current | 3
  Former | 26
  Never | 6
Baseline ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; and 5=Dead.
  Participants
    ECOG = 1 | 26
    ECOG = 0 | 9
Prior checkpoints inhibitors (CPI) [Count of Participants; unit: Participants]
  Pembrolizumab | 21
  Nivolumab | 7
  Atezolizumab | 5
  Durvalumab | 1
  Spartalizumab | 1
First-line Chemo [Count of Participants; unit: Participants]
  Carboplatin + Pemetrexed | 21
  Carboplatin + Taxane | 12
  Cisplatin based chemo | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progressive Disease (PD): >= 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  PFS was defined as time from starting treatment to disease progression met by RECIST 1.1, start of additional anticancer therapy before progression, or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 35
months | 5.1 [3.6 to 8]

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Per Immune-Related RECIST (irRECIST): Complete Response(irCR), Disappearance of all measurable and non-measurable lesions; Partial Response (irPR) >=30% decrease in tumor burden relative to baseline; Progressive Disease (irPD), >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions confirmed by a consecutive assessment at least 4 week after first documentation; Stable Disease (irSD), not meeting criteria for irCR or irPR, in absence of irPD CBR is defined as any subject with SD for ≥ 3 months, PR or CR assessed via RECIST 1.1 and irRECIST.
Time Frame: Up to a maximum of 28 months
Population: Out of 35 patients in the study, one subject was not evaluable for best response using RECIST 1.1 and two subjects were not evaluable for best response using irRECIST.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 34
Participants
  CBR by RECIST1.1 | 24
  CBR by irRECIST: number analyzed (Participants) | 33
  CBR by irRECIST | 24

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Per RECIST: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Per irRECIST: Complete Response(irCR), Disappearance of all measurable and non-measurable lesions; Partial Response (irPR) >=30% decrease in tumor burden relative to baseline; Progressive Disease (irPD), >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions confirmed by a consecutive assessment at least 4 week after first documentation; Stable Disease (irSD), not meeting criteria for irCR or irPR, in absence of irPD ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1 and irRECIST, from the start of treatment until disease progression/recurrence
Time Frame: Up to a maximum of 28 months
Population: Out of 35 patients, one subject was not evaluable for best response using RECIST 1.1 and two subjects were not evaluable for best response using irRECIST.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 34
percentage of participants
  ORR by RECIST1.1 | 23.5 [10.8 to 41.2]
  ORR by irRECIST: number analyzed (Participants) | 33
  ORR by irRECIST | 27.3 [13.3 to 45.5]

4. Secondary Outcome: Overall Survival (OS)
Description: Time from date of treatment start to date of death from any cause
Time Frame: Time of treatment start until death or up to a maximum of 40 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 35
months | 24.5 [15.6 to 30.9]

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicity will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 4
Time Frame: Adverse events were recorded from time of registration until 30 days after discontinuation of study drug(s) up to a maximum of 25 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 35
Participants | 35

6. Secondary Outcome: Progression Free Survival (PFS) by irRECIST
Description: Per Immune-Related RECIST (irRECIST): Complete Response(irCR), Disappearance of all measurable and non-measurable lesions; Partial Reponse (irPR): >=30% decrease in in tumor burden relative to baseline; Progressive Disease (irPD), >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions confirmed by a consecutive assessment at least 4 week after first documentation; Stable Disease (irSD), not meeting criteria for irCR or irPR, in absence of irPD.
  PFS is defined as time from the date of treatment start until the criteria for disease progression is met as defined by irRECIST or death occurs.
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
Number analyzed (Participants) | 35
months | 5.2 [3.6 to 9.8]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 40 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored from the initiation of study therapy until 30 days after treatment discontinuation, up to 25 months.
Arm/Group | Pembrolizumab 200mg IV Every 21 Days
All-Cause Mortality (participants affected / at risk) | 18/35
Serious Adverse Events (participants affected / at risk) | 11/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200mg IV Every 21 Days (N=35)
ANEMIA (Blood and lymphatic system disorders) | 2 (2)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FEVER (General disorders) | 2 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200mg IV Every 21 Days (N=35)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6 (15)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 8 (10)
ALOPECIA (Skin and subcutaneous tissue disorders) | 7 (9)
AMNESIA (Nervous system disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 22 (86)
ANOREXIA (Metabolism and nutrition disorders) | 14 (19)
ANXIETY (Psychiatric disorders) | 13 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (6)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 8 (13)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (17)
BLADDER INFECTION (Infections and infestations) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (3)
BLURRED VISION (Eye disorders) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 1 (3)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 2 (2)
CD4 LYMPHOCYTES DECREASED (Investigations) | 2 (3)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 5 (6)
CHILLS (General disorders) | 3 (3)
CHOLESTEROL HIGH (Investigations) | 10 (10)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 (1)
CONFUSION (Psychiatric disorders) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 15 (19)
COUGH (Respiratory, thoracic and mediastinal disorders) | 27 (39)
CREATININE INCREASED (Investigations) | 8 (18)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4)
DEPRESSION (Psychiatric disorders) | 13 (15)
DIARRHEA (Gastrointestinal disorders) | 11 (24)
DIZZINESS (Nervous system disorders) | 7 (9)
DRY EYE (Eye disorders) | 4 (4)
DRY MOUTH (Gastrointestinal disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3)
DYSESTHESIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 7 (9)
DYSPEPSIA (Gastrointestinal disorders) | 3 (4)
DYSPHAGIA (Gastrointestinal disorders) | 2 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 24 (42)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 1 (2)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA FACE (General disorders) | 1 (3)
EDEMA LIMBS (General disorders) | 16 (32)
EDEMA TRUNK (General disorders) | 1 (2)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (5)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 8 (10)
FALL (Injury, poisoning and procedural complications) | 3 (3)
FATIGUE (General disorders) | 26 (73)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
FEVER (General disorders) | 10 (19)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
FLU LIKE SYMPTOMS (General disorders) | 1 (1)
FLUSHING (Vascular disorders) | 2 (2)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (2)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 2 (5)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 11 (12)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 4 (4)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 8 (10)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 9 (12)
HEARING IMPAIRED (Ear and labyrinth disorders) | 2 (2)
HEART FAILURE (Cardiac disorders) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (3)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HOT FLASHES (Vascular disorders) | 3 (3)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPERTENSION (Vascular disorders) | 20 (49)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 5 (12)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 10 (22)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 3 (4)
HYPOTHYROIDISM (Endocrine disorders) | 10 (10)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (3)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 4 (4)
INFUSION RELATED REACTION (General disorders) | 2 (3)
INSOMNIA (Psychiatric disorders) | 15 (17)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 2 (2)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1)
LOCALIZED EDEMA (General disorders) | 4 (5)
LUNG INFECTION (Infections and infestations) | 2 (2)
LYMPH GLAND INFECTION (Infections and infestations) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1)
MALAISE (General disorders) | 2 (2)
MUCOSITIS ORAL (Gastrointestinal disorders) | 5 (7)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 8 (8)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (8)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 2 (3)
NAIL INFECTION (Infections and infestations) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 8 (13)
NAUSEA (Gastrointestinal disorders) | 21 (68)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 (11)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 12 (43)
NON-CARDIAC CHEST PAIN (General disorders) | 5 (7)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN (General disorders) | 11 (21)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (12)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 4 (4)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 10 (17)
PHARYNGEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PHLEBITIS (Vascular disorders) | 3 (4)
PLATELET COUNT DECREASED (Investigations) | 7 (27)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 (7)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 4 (4)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 9 (19)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 13 (31)
RECTAL MUCOSITIS (Gastrointestinal disorders) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 12 (13)
RHINITIS INFECTIVE (Infections and infestations) | 1 (1)
SCLERAL DISORDER (Eye disorders) | 1 (1)
SINUS PAIN (Nervous system disorders) | 1 (1)
SINUSITIS (Infections and infestations) | 3 (5)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 6 (7)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (3)
SKIN INFECTION (Infections and infestations) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 2 (3)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 2 (3)
SYNCOPE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 4 (6)
TOOTH INFECTION (Infections and infestations) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 5 (8)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 3 (5)
URINARY URGENCY (Renal and urinary disorders) | 1 (1)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1)
VAGINAL INFLAMMATION (Reproductive system and breast disorders) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 2 (4)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 13 (26)
WATERING EYES (Eye disorders) | 4 (4)
WEIGHT GAIN (Investigations) | 9 (14)
WEIGHT LOSS (Investigations) | 3 (8)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 5 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03083808/Prot_SAP_001.pdf